CLINICAL TRIAL: NCT02603783
Title: "Effect of capsaïcin Infusion on Esophageal Mucosal Integrity - a Role for TRPV1-mediated Neuropeptides?"
Brief Title: Esophageal capsaïcin Infusion and Mucosal Integrity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: METC 152005
Record Dates: First submitted 2015-10-30; First posted 2015-11-13 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2015-10

CONDITIONS: TRPV1 Protein, Human; Capsaicin; Electric Impedance; Esophagus; Intracellular Space; Pain Measurement; Microscopy, Electron
MeSH Terms: interventions — Capsaicin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capsaicin (Active Comparator): 1,5 mg capsaicin in 30 minutes
  Interventions: Other: Capsaicin
- Placebo (Placebo Comparator): 75 ml placebo (0,9 % saline) in 30 minutes
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Capsaicin — capsaicin 1,5 mg
  Arms: Capsaicin
Other: Placebo — 0,9% saline 75 ml
  Arms: Placebo

SUMMARY:
Reflux is common, especially after large meals. In general, this can do no harm. However, if reflux occurs often and causes troublesome symptoms and or complications, it is called gastroesophageal reflux disease (GERD). Long exposure to gastric acid causes the mucosa of the esophagus to loose its integrity, which is thought to lead to the symptom of heartburn. Several food products can also impair the esophageal mucosa integrity and thereby influence reflux symptoms. One of these products is capsaicin, the pungent ingredient of red peppers. Use of capsaicin often leads to worsening of complaints in patients with GERD and can cause symptoms in healthy volunteers, possibly due to its effect on the mucosal integrity.

In this study the investigators want to investigate the effect of capsaicin infusion on mucosal integrity. The investigators will evaluate mucosal impedance and the histology of the esophageal mucosa. In addition, the investigators also aim to assess the involvement of the TRPV1 receptor by evaluating the possible release of neuropeptides in the esophageal mucosa.

ELIGIBILITY:
Inclusion Criteria:

* No history of gastrointestinal disease, especially gastro-esophageal reflux disease.
* BMI = 18-25 kg/m²
* Caucasian race
* Subject signed the informed consent form and is able to adhere to study protocol

Exclusion Criteria:

* Age <18 years
* Erosive esophagitis or gastric ulceration during endoscopy on PPI in the past or during the experiment
* Use of regular (> 1 x per week) dietary capsaïcin (in additives as Tabasco/sambal/chili sauce or Indian, Mexican or Thai food dishes)
* Allergy to capsaïcin
* Use of medication affecting GI function (prokinetics) or antisecretory medication (PPI) within 3 days prior to endoscopy.
* Multisystem diseases (including severe cardiopulmonary disease, collagen diseases, coagulation disorders)
* Esophageal motility disorders
* Previous esophageal or gastric surgery
* Use of anticoagulants or a history of coagulopathy
* Pregnancy
* History of alcohol abuse or current excessive alcohol consumption (> 2 alcoholic beverages per day or > 14 alcoholic beverages per week)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-11; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Changes in mucosal integrity in the distal exposed esophagus during capsaicin infusion compared to control solution. | Testday 1 and 2: mucosal biopsies are taken during upper gastrointestinal endoscopy
  The primary outcome measure is the effect of capsaïcin infusion on mucosal integrity as reflected by baseline impedance in the distal exposed esophagus compared to control infusion.
  We hypothesize that capsaïcin infusion induces changes to the mucosa as reflected by a decrease in baseline impedance.

SECONDARY OUTCOMES:
Mucosal integrity in the proximal non-exposed esophagus. | Testday 1 and 2: mucosal biopsies are taken during upper gastrointestinal endoscopy
  The effect of esophageal capsaïcin infusion on mucosal integrity as reflected by baseline impedance in the proximal non-exposed esophagus compared to control solution.
Induction of dilated intercellular spaces (DIS) | Testday 1 and 2: mucosal biopsies are taken during upper gastrointestinal endoscopy
  The effect of esophageal capsaïcin infusion on the induction of dilated intercellular spaces (DIS) in the distal exposed and proximal non-exposed esophagus as measured with transmission electron microscopy (TEM).
TRPV1 neuropeptide pathway | Testday 1 and 2: mucosal biopsies are taken during upper gastrointestinal endoscopy
  The differences in the TRPV1 neuropeptide pathway (substance P) by radioimmunoassay (RIA) during capsaïcin infusion or control solution in both the distal exposed and proximal non-exposed esophagus.
Immunohistochemical expression of TRPV1 | Testday 1 and 2: mucosal biopsies are taken during upper gastrointestinal endoscopy
  The differences in immunohistochemical expression of TRPV1 during capsaïcin infusion or control solution in both the distal exposed and proximal non-exposed esophagus.
Symptom scores | Testday 1 and 2: during capsaicin and placebo infusion.
  The effect of capsaïcin infusion on symptoms in healthy volunteers.
TRPV1 neuropeptide pathway | Testday 1 and 2: mucosal biopsies are taken during upper gastrointestinal endoscopy
  The differences in the TRPV1 neuropeptide pathway (CGRP) by radioimmunoassay (RIA) during capsaïcin infusion or control solution in both the distal exposed and proximal non-exposed esophagus.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Conchillo, MD, PhD, Principal Investigator — Maastricht University Medical Center (MUMC+)
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Alleleyn AME, Keszthelyi D, Rinsma NF, Cseko K, Kajtar B, Helyes Z, Winkens B, Masclee AAM, Conchillo JM. The Potential Role for Impaired Mucosal Integrity in the Generation of Esophageal Pain Using Capsaicin in Humans: An Explorative Study. Clin Transl Gastroenterol. 2022 May 1;13(5):e00488. doi: 10.14309/ctg.0000000000000488. PMID 35351835